CLINICAL TRIAL: NCT07107789
Title: The Effect of Diabetes Education Delivered Through Video Animation on Metabolic Control, Self-Care Ability, Perceived Social Support, and Attitudes Toward the Disease in Children With Type 1 Diabetes
Brief Title: The Effect of Diabetes Education Given With Video Animation on Metabolic Control, Self-Care Ability, and Attitudes Towards the Disease in Children With Type 1 Diabetes
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Gamze Nur Yılmaz, Phd Student, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: AU-SBE-GNY-01
Record Dates: First submitted 2025-07-11; First posted 2025-08-06 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-07

CONDITIONS: Type 1 Diabetes in Children
Keywords: child; diabetes; animation; education; metabolic; control; self-care
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: Two groups, the traditional experimental and control groups
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The control group will receive routine diabetes education from the hospital's diabetes nurse. The experimental group will receive diabetes education using a video animation prepared by the researcher following the routine diabetes education provided by the diabetes nurse. The outcome assessment and group allocation will be conducted by a researcher who is unaware of the outcome.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The experimental group will receive diabetes education through video animation. (Active Comparator): Following the routine diabetes education provided by the hospital, the experimental group will receive diabetes education using a video animation prepared by the researcher and approved by an expert. Pre- and post-intervention surveys will be administered.
  Interventions: Other: Diabetes education with video animation
- Control group to receive routine diabetes education (No Intervention): The control group will receive routine diabetes education from the hospital's diabetes nurse. No intervention will be applied. Only the scale and pre-test/post-test will be administered to the control groups.

INTERVENTIONS:
Other: Diabetes education with video animation — Providing diabetes education to the experimental group through a video animation Following the routine diabetes education provided by the hospital, the experimental group will receive diabetes education using a video animation prepared and staged by the researcher and approved by experts.
  Arms: The experimental group will receive diabetes education through video animation.

SUMMARY:
The aim of this study is to evaluate the attitude towards the disease, perceived social support systems, metabolic control and self-care ability of pediatric patients diagnosed with Type 1 diabetes, by giving video animation training considering their age and developmental level. The main questions it aims to answer are:

1. Nursing interventions using video animations increase self-care abilities in children aged 11-18.
2. Nursing interventions using video animations increase the perception of social support in children aged 11-18.
3. Nursing interventions using video animations support metabolic control in children aged 11-18.
4. Nursing interventions using video animations positively affect the attitudes of children aged 11-18 toward their illness.

DETAILED DESCRIPTION:
With the development and proliferation of technology, an essential part of our daily lives, adaptation and developments in technology have begun to increase in the healthcare sector. Research has shown that games and video animations are effective methods beyond medication. No studies have been found in the literature evaluating the effects of diabetes education provided through video animation on the metabolic control, self-care abilities, and attitudes toward the disease in children with Type 1 diabetes. Therefore, the aim of this study is to evaluate the effects of video animation education given to children diagnosed with Type 1 diabetes on their attitudes toward the disease, perception of social support, and self-care abilities. It is anticipated that this research will provide a proactive, multifaceted approach to care and treatment. The study was designed as a pretest/posttest randomized controlled trial. The study population consisted of children aged 11-18 who were regularly followed in the outpatient clinic and had been diagnosed with Type 1 diabetes for at least 6 months. Children who accepted the study and met the criteria were assigned to the video animation and control groups using a block randomization method. The study sample was determined to be 80 individuals, 40 in the experimental group and 40 in the control group. The video animation scenario to be used in the study was created by the researchers in parallel with the routine diabetes education provided at the hospital, and expert approval was obtained. The video animation scenes were prepared by a voice actor and illustrator as part of the project. The experimental group will receive diabetes education through video animation following the routine diabetes education provided by the hospital. Pre- and post-intervention surveys will be administered. The control group will receive routine diabetes education from the hospital's diabetes nurse. No other intervention will be administered. Pre-tests/post-tests and surveys will be administered before and after the diabetes education.

ELIGIBILITY:
Inclusion Criteria:

* Agreeing to participate in the study
* Diagnosed with Type 1 DM by a specialist
* Diagnosed with Type 1 diabetes for at least 6 months
* Being between the ages of 11 and 18
* Using an insulin pen
* Not using an insulin pump
* Coming for regular checkups at the Pediatric Endocrinology clinic
* Having no other chronic disease besides diabetes

Exclusion Criteria:

* Using an insulin pump
* Not being mentally healthy
* Having any mental or physical disability

Ages: 11 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-08-15 (Estimated); Primary Completion 2025-09-15 (Estimated); Study Completion 2025-10-06 (Estimated)

PRIMARY OUTCOMES:
Metabolic Control | three weeks
  Weight and height measurements will be combined to report body mass index in kg/m². Fasting and postprandial blood glucose values and HbA1C values will be evaluated.
Self-care power | three weeks
  The five-point Likert-type self-care agency scale, which offers an opportunity for self-assessment, consists of 35 questions. The total score obtained from the scale ranges from 35 to 140. A higher total score indicates that the patient is more independent and competent in self-care.
Attitude Towards One's Own Illness | three weeks
  It provides an opportunity to assess the attitudes children with chronic illness develop toward their illness. A 13-item, five-point Likert-type scale was designed to self-report children with chronic illnesses. Four of the 13 items are bipolar (very good, somewhat good, not sure, somewhat bad, very bad), while nine items assess how often children experience positive or negative feelings specific to having a chronic illness, using the phrases "very often, often, sometimes, not often, never." Mean scores for items measuring children's attitudes toward their illnesses range from 1 to 5. The lowest possible total score is 13, and the highest is 65. There are no reverse items. Scores of 1 and 2 indicate a negative attitude, 3 indicate a neutral attitude, and 4 and 5 indicate a positive attitude. The internal consistency coefficient of the scale was determined to be 0.79.
Multifaceted Perceived Social Support | three weeks
  The total score available ranges from 12 to 84. A higher score indicates a positive perception of social support.

CONTACTS AND LOCATIONS:
Overall Officials: Gamze Nur YILMAZ, PhD, Principal Investigator — Ataturk University
Locations (1):
- Erzurum City Hospital, Erzurum, Palandöken, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No